CLINICAL TRIAL: NCT00115947
Title: Renal and Cardiovascular Effects of Terlipressin in Patients With Cirrhosis and Ascites
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2004-000568-29
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2006-03-09 (Estimated); Status verified 2005-06

CONDITIONS: Cirrhosis; Ascites
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Terlipressin

INTERVENTIONS:
Drug: Terlipressin

SUMMARY:
The purpose of this study is to investigate the effect of terlipressin on myocardial perfusion and renal function.

Hypothesis: Significant improvement of renal function reflected by: glomerular filtration rate (GFR), renal blood flow (RBF), excretion of salt and metabolites in the urine and related hormones and peptides in the blood. No effect on the systolic function of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis and ascites

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Krag Krag, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Copenhagen, Hvidovre, Denmark